CLINICAL TRIAL: NCT00992173
Title: A Phase 2b Study Evaluating the Efficacy and Safety of Ultratrace™ Iobenguane I 131 Among Patients With Relapsed/Refractory High-Risk Neuroblastoma
Brief Title: Efficacy and Safety of Ultratrace™ Iobenguane I 131 in Neuroblastoma
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Molecular Insight Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MIP-IB-N201
Record Dates: First submitted 2009-10-07; First posted 2009-10-09 (Estimated); Last update posted 2015-11-26 (Estimated); Status verified 2015-11

CONDITIONS: Neuroblastoma
Keywords: Neuroblastoma; MIBG; Iobenguane
MeSH Terms: conditions — Neuroblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ultratrace Iobenguane I 131 (Experimental)
  Interventions: Drug: Ultratrace Iobenguane I 131

INTERVENTIONS:
Drug: Ultratrace Iobenguane I 131 — Subjects will receive an Imaging Dose of 0.1 mCi/kg [3.7 MBq/kg] (a minimum dose of 1.0 mCi [37 MBq] but not to exceed 5.0 mCi [185 MBq]) of Ultratrace iobenguane I 131 to have dosimetry performed and to confirm tumor uptake of the test article prior to receiving each of 2 planned Therapeutic Doses of Ultratrace iobeneguane I 131 . Within 28 days of screening, eligible subjects (as confirmed by the first Imaging dose study)will receive an Ultratrace iobenguane I 131 Therapeutic dose of of 15.0 - 18.0 mCi/kg (max. 666 MBq/kg) followed by imaging 7 days later or upon discharge from radiation isolation. A second Therapeutic Dose (preceded by a repeat Image Dose and dosimetry study)and imaging upon discharge from radiation isolation will be repeated approximately 8 weeks after the first dose.

SUMMARY:
This is a multi-center, single arm trial of two doses of 18 mCi/kg of Ultratrace iobenguane I 131 administered to subjects with high-risk neuroblastoma. Iobenguane I 131 is a drug that has already been used in many children to treat neuroblastoma, and it is known to shrink some of the tumors, and cause manageable side effects. When administered intravenously, Iobenguane I 131 accumulates in the neuroblastoma cancer cells and causes them to die.

In this study the investigators are investigating the use of a new form of Iobenguane I 131 called Ultratrace iobenguane I 131. This form is expected to deliver higher amounts of radioactive I 131 to the neuroblastoma cells. The primary purpose of the study is to determine if Ultratrace iobenguane I 131 can be used to successfully treat high-risk neuroblastoma. The study will also assess the safety of Ultratrace iobenguane I 131 when given to patients with high-risk neuroblastoma.

ELIGIBILITY:
Patients must meet all of the following inclusion criteria:

1. Males or females who are >12 months of age
2. Have a diagnosis of neuroblastoma either by (a) histologic verification of neuroblastoma and/or (b) demonstration of tumor cells in the bone marrow with increased urinary catecholamine metabolites
3. Have high-risk neuroblastoma with relapsed/refractory disease at any time.
4. MIBG avid disease demonstrated by 131I or 123I -MIBG uptake into tumor at ≥ one site within 28 days prior to study treatment and no intervention/therapy between the time of the MIBG scan and study treatment.
5. To be eligible to receive at least one therapeutic dose, patients must have adequate banked autologous stem cells defined as:

   PBSC: A minimum of 2.0 x 106 viable CD34+ cells/kg (purged or unpurged) (see Section 10.4.15)
6. Prior Therapy:

   1. Patients must have fully recovered from the acute toxic effects of all prior chemotherapy, immunotherapy, or radiotherapy prior to entering this study. There is no limitation on the number of prior chemotherapeutic regimens that the patient may have received.
   2. The last dose of all local palliative radiation must be ≥ 14 days prior to the first therapeutic dose of Ultratrace iobenguane I 131. Any lesion treated with local palliative radiation during this period can not be included in the baseline target lesion evaluation.
   3. The last dose of all local palliative radiation to more than 25% of marrow containing bones must be ≥ 28 days prior to the first therapeutic dose of Ultratrace iobenguane I 131. A minimum of 3 months is required following prior large field radiation therapy (i.e. craniospinal therapy, total lung, > 50% marrow space). Note: Radiation therapy of focal skull-based bony metastatic disease (only) is not considered craniospinal therapy.
   4. The last dose of any myelosuppressive or biologic (e.g., isotretinoin [also known as cis-retinoic acid, or Accutane®]) therapy must be at least 14 days before the administration of the first therapeutic dose of Ultratrace iobenguane I 131 on this protocol.
   5. The last dose of immunotherapy must be at least 28 days prior to the first therapeutic dose of Ultratrace iobenguane I 131.
   6. All cytokines or hematopoietic growth factors must be discontinued for a minimum of 7 days prior to the first therapeutic dose of Ultratrace iobenguane I 131or 14 days prior to the first therapeutic dose of Ultratrace iobenguane I 131for long-acting colony stimulating factors.
   7. Prior treatment with 131I-MIBG therapy must be ≥12 months prior to the first therapeutic dose of Ultratrace iobenguane I 131.
   8. Administration of Neuroblastoma therapeutic investigational medication or devices must be ≥30 days prior to dosimetry dose.
   9. Prior autologous stem cell infusion must be ≥2 months prior to study entry. The patient must have recovered from all toxicities
7. Adequate Organ Function:

   1. Adequate bone marrow function requirements, including patients post-myeloablative therapy or tumor involvement of bone marrow
   2. Adequate renal, hepatic, cardiac, lung and thyroid function

Exclusion Criteria:

Patients will be excluded if any of the following conditions are observed:

1. Pregnant, or lactating females with the intent to breast feed. Females of child-bearing potential must have a negative serum pregnancy test prior to therapy. Males and females of reproductive age and childbearing potential must use effective contraception defined as abstinence or use of IUD, oral contraceptive, barrier and spermicide, or hormonal implant for the duration of their participation. Sexually active female patients using oral contraception will be required to use a second form of barrier birth control. All patients will be required to use effective contraception for 60 days following the last therapeutic dose of Ultratrace iobenguane I 131.
2. Have disease of any major organ system that would compromise their ability to withstand therapy.
3. Receiving hemodialysis or have a renal obstruction, which would effect the urinary excretion of MIBG.
4. Is platelet transfusion dependent
5. Status post-allogeneic hematopoietic stem cell transplant.
6. Concomitant use of medications that inhibit uptake of Ultratrace iobenguane I 131.
7. Have a known allergy to iobenguane, iodine or SSKI.
8. If patients and/or families who are physically and psychologically unable to cooperate with the radiation safety isolation or imaging requirements (sedation or general anesthesia permitted).
9. Administered prior chemotherapy within 30 days of study entry or have active malignancy (other than neuroblastoma) requiring additional treatment.
10. Any other condition, that in the opinion of the investigator, may compromise the safety or compliance of the subject or would preclude the subject from successful completion of the study.
11. Patient unable to receive at least one 15 mCi/kg dose per dosimetry findings.

Min Age: 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-01; Primary Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with complete or partial response, sustained over two assessments, following treatment. Response criteria for the primary endpoint are based on the International Neuroblastoma Response Criteria (INRC). | Weeks 8, 16, 26, 39 and 52 after treatment

SECONDARY OUTCOMES:
Change in use of narcotics for pain management | Weeks 8, 16, 26, 39 and 52 after treatment
Change in patient quality of life | Weeks 8, 16, 26, 39 and 52 after treatment
Change in key tumor markers (HVA and VMA) | Weeks 8, 16, 26, 39 and 52 after treatment
Overall survival | Weeks 8, 16, 26, 39 and 52 after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Norman LaFrance, MD, Study Director — Molecular Insight Pharmaceutical Employee
Locations (21):
- United States (20):
  - Children's Hospital of LA, Los Angeles, California
  - UCSF Pediatric Hematology/Oncology, San Francisco, California
  - University of Miami Miller School of Medicine, Miami, Florida
  - Childrens Memorial/Northwestern University, Chicago, Illinois
  - Comer's Childrens Hospital/University of Chicago, Chicago, Illinois
  - University of iowa, Iowa City, Iowa
  - Johns Hopkins University, Baltimore, Maryland
  - Children's Hospital/Dana Farber Cancer Institute, Boston, Massachusetts
  - CS Motts Children's Hospital, Ann Arbor, Michigan
  - Mount Sinai School of Medicine, New York, New York
  - Hospital - Weill Cornell Medical Center, New York, New York
  - Memorial Sloan Kettering, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Cook Children's Healthcare System, Fort Worth, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - Texas Childrens Hospital Cancer Center, Houston, Texas
  - University of Wisconsin Medical Center, Madison, Wisconsin
- The Hospital for Sick Children, Toronto, Ontario, Canada